CLINICAL TRIAL: NCT04212806
Title: French Linguistic Validation of Questionnaires for Patients With Axial Spondyloarthritis
Brief Title: French Validation of Axial Spondyloarthritis Questionnaires (Val-SpA)
Acronym: Val-SpA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.291; 2019-A02508-49 (Other: ID RCB)
Record Dates: First submitted 2019-11-25; First posted 2019-12-30 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis
Keywords: Validation; BASFI; Dougados Functional Index; BAS-G
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to do a French linguistic validation of three questionnaires used in axial Spondyloarthritis (BASFI, BAS-G, Dougados Functional Index).

In order to validate the questionnaires, a prospective, qualitative, observational and monocentric study will be conducted.

DETAILED DESCRIPTION:
Axial spondyloarthritis (SpA) is a chronic rheumatic diseases affecting axial skeleton and sacro-iliac joints. SpA can have functional consequences, often assessed with the Bath Ankylosing Spondylitis Functional Index (BASFI), the Dougados functional index, or more globally with the Bath Ankylosing Spondylitis Global (BAS-G). If these questionnaires are validated in English, there are not validated in French. The aim is to do a french linguistic validation of these questionnaires.

A translation, reconciliation and retro-translation will be conducted for each of the questionnaires by two bilingual translators. The last version of each questionnaire will be then validated by clinicians experts in SpA. The version will be further validated by 5 patients. If necessary and if changes occured on the version of the questionnaire, another version will be validated by 5 other patients until full understanding is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with axial spondyloarthritis or ankylosing spondylitis

Exclusion Criteria:

* Patients who do not understand French
* Patients with cognitive impairments
* People protected by law
* People who do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Ankylosing Spondylitis or Axial Spondyloarthritis at any stage of disease evolution followed at the Rhumatology unit of Grenoble University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
BASFI validity in French | Day 0
  The self-administered Bath Ankylosing Spondylitis Functional Index (BASFI) measures functional consequences of axial spondyloarthritis. The score will be validated in French if the clarity and understanding is approved by 5 french native-language patients.
BAS-G validity in French | Day 0
  The self-administered Bath Ankylosing Spondylitis Global (BAS-G) measures global consequences of axial spondyloarthritis on well-being. The score will be validated in French if the clarity and understanding is approved by 5 french native-language patients.
Dougados validity in French | Day 0
  The self-administered Dougados functional Index measures functional capacities of patients with axial spondyloarthritis. The score will be validated in French if the clarity and understanding is approved by 5 french native-language patients.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Grenoble Alpes, Grenoble
  - CHU Grenoble Alpes, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soulard J, Vaillant J, Baillet A, Vuillerme N. Translation and French Linguistic Validation of the Bath Ankylosing Spondylitis Functional Index and the Bath Ankylosing Spondylitis Global Score in Patients with Axial Spondyloarthritis. Curr Rheumatol Rev. 2023;19(4):449-454. doi: 10.2174/1573397118666220829124234. PMID 36043728